CLINICAL TRIAL: NCT02257398
Title: A Phase I, Randomized, Double-Blinded, Placebo- and Moxifloxacin-Controlled, 4-Period Crossover Study to Evaluate the Effect of GSK2140944 on Cardiac Conduction as Assessed by 12-lead Electrocardiogram in Healthy Volunteers
Brief Title: Placebo and Moxifloxacin Controlled Cardiac Conduction Study of GSK2140944 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 115775
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Infections, Respiratory Tract
Keywords: TQTc; Moxifloxacin; GSK2140944
MeSH Terms: conditions — Respiratory Tract Infections | interventions — gepotidacin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence ABDC (Experimental): Subjects will be administered treatments in Sequence ABDC where, A= GSK2140944 1000 mg IV infusion over 120 minutes and single dose of moxifloxacin placebo administered orally in morning; B= GSK2140944 1800 mg IV infusion over 120 minutes and single dose of moxifloxacin placebo administered orally in morning; C= GSK2140944 placebo IV infusion over 120 minutes and single dose of moxifloxacin placebo administered orally in morning and D= Moxifloxacin 400 mg administered orally in morning and GSK2140944 placebo administered as IV infusion over 120 minutes
  Interventions: Drug: GSK2140944; Drug: GSK2140944 placebo; Drug: Moxifloxacin; Drug: Moxifloxacin placebo
- Sequence BCAD (Experimental): Subjects will be administered treatments in Sequence BCAD where, A= GSK2140944 1000 mg IV infusion over 120 minutes and single dose of moxifloxacin placebo administered orally in morning; B= GSK2140944 1800 mg IV infusion over 120 minutes and single dose of moxifloxacin placebo administered orally in morning; C= GSK2140944 placebo IV infusion over 120 minutes and single dose of moxifloxacin placebo administered orally in morning and D= Moxifloxacin 400 mg administered orally in morning and GSK2140944 placebo administered as IV infusion over 120 minutes
  Interventions: Drug: GSK2140944; Drug: GSK2140944 placebo; Drug: Moxifloxacin; Drug: Moxifloxacin placebo
- Sequence CDBA (Experimental): Subjects will be administered treatments in Sequence CDBA where, A= GSK2140944 1000 mg IV infusion over 120 minutes and single dose of moxifloxacin placebo administered orally in morning; B= GSK2140944 1800 mg IV infusion over 120 minutes and single dose of moxifloxacin placebo administered orally in morning; C= GSK2140944 placebo IV infusion over 120 minutes and single dose of moxifloxacin placebo administered orally in morning and D= Moxifloxacin 400 mg administered orally in morning and GSK2140944 placebo administered as IV infusion over 120 minutes
  Interventions: Drug: GSK2140944; Drug: GSK2140944 placebo; Drug: Moxifloxacin; Drug: Moxifloxacin placebo
- Sequence DACB (Experimental): Subjects will be administered treatments in Sequence DACB where, A= GSK2140944 1000 mg IV infusion over 120 minutes and single dose of moxifloxacin placebo administered orally in morning; B= GSK2140944 1800 mg IV infusion over 120 minutes and single dose of moxifloxacin placebo administered orally in morning; C= GSK2140944 placebo IV infusion over 120 minutes and single dose of moxifloxacin placebo administered orally in morning and D= Moxifloxacin 400 mg administered orally in morning and GSK2140944 placebo administered as IV infusion over 120 minutes
  Interventions: Drug: GSK2140944; Drug: GSK2140944 placebo; Drug: Moxifloxacin; Drug: Moxifloxacin placebo

INTERVENTIONS:
Drug: GSK2140944 — GSK2140944 is available in dose strength 1000 mg and 1800 mg for single IV dose over 2 hours administration as a pale yellow to greyish yellow cake for reconstitution
Drug: GSK2140944 placebo — GSK2140944 placebo is 0.9% sodium chloride available for single IV dose over 2 hours administration.
Drug: Moxifloxacin — Moxifloxacin is available as pinkish red tablet with dose strength 400 mg for single oral dose to be administered in the morning in the fasted state with approximately 240 mL of water.
Drug: Moxifloxacin placebo — Moxifloxacin placebo is available as white, film-coated tablet. containing nonactive material for single oral dose to be administered in the morning in the fasted state with approximately 240 mL of water.

SUMMARY:
This is Phase I, 4-period, randomized, active-and placebo-controlled, double-blind crossover, single-dose study to evaluate the effects of a therapeutic (1000 milligram [mg]) and supratherapeutic (1800 mg) dose of GSK2140944 with a positive control (moxifloxacin 400 mg) and placebo on the corrected QT interval (QTc) as assessed by continuous 12-lead Holter electrocardiograms (ECGs) in approximately 55 healthy volunteers.

All subjects will receive single doses of GSK2140944 1000 mg, GSK2140944 1800 mg, moxifloxacin 400 mg, and placebo in a randomized sequence. A double-dummy approach will be used to maintain blinding. Thus, on each dosing day, moxifloxacin or moxifloxacin placebo and GSK2140944 or placebo will be administered.

Subjects will be screened within 30 days prior to entry to the clinic. Subjects will report to the clinical unit on Day -2 of Period 1 and on Day -1 in subsequent periods. Subjects will remain confined until check out procedures have been completed on Day 3 (5 days confinement in Period 1 and 4 days in the following 3 periods). There will be a washout of at least 7 days between doses. The follow-up visit will occur 7-10 days after the final dose. Total duration of the study (from screening to the follow-up visit) will be approximately 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 55 years of age, inclusive, at the time of signing the informed consent
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the investigator feels and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >= 50 kilogram (kg) and body mass index within the range 19 to 31 kilogram / square meter (kg/m^2) (inclusive).
* A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum beta-human chorionic gonadotrophin test), not lactating, and at least one of the following conditions applies:
* Nonreproductive potential defined as:
* Premenopausal females with one of the following: Documented tubal ligation, documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, hysterectomy, documented bilateral oophorectomy.
* Postmenopausal defined as 12 months of spontaneous amenorrhea. To confirm postmenopausal status, a blood sample for simultaneous follicle-stimulating hormone (FSH) >40 milli-international units per mililiter (mlU/mL) and estradiol <40 picogram/milliliter (pg/mL) (<147 picomole/liter [pmol/L]) is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status prior to study enrolment.
* Reproductive potential and agrees to follow one of the options listed below in the GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) requirements from 30 days prior to the first dose of study drug and until at least 7 days after the last dose of study drug and completion of the follow-up visit.
* This list does not apply to FRP with same sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penile-vaginal intercourse on a long-term and persistent basis.
* Contraceptive subdermal implant that meets the standard operating procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label, intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label, oral contraceptive, either combined or progestogen alone, injectable progestogen, contraceptive vaginal ring, percutaneous contraceptive patches, male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject.
* These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Capable of giving signed informed consent as described in protocol, which includes compliance with the requirements and restrictions listed in the consent form and in the protocol
* Alanine aminotransferase (ALT) and bilirubin <1.5 × upper limit of normal range (ULN). Isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%. One repeat test to confirm result is acceptable.
* Serum potassium, calcium, and magnesium laboratory parameters within normal limits at screening and check-in.

Exclusion Criteria:

* History/evidence of any arrhythmia (for example, second- or third-degree heart block, atrial fibrillation, supraventricular tachycardia, symptomatic sinus bradycardia, junctional rhythm) or clinically significant cardiac disease or procedure (mitral valve regurgitation, heart murmur, angina/ischemia, congenital heart abnormalities, coronary artery bypass grafting surgery, or percutaneous transluminal coronary angioplasty). A history of additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia, and family history of long QT syndrome).
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert syndrome or asymptomatic gallstones).
* Any clinically significant CNS (e.g., seizures), cardiac, pulmonary, metabolic, renal, hepatic, or GI conditions or history of such conditions that, in the opinion of the investigator, may place the subject at an unacceptable risk as a participant in this trial or may interfere with the absorption, distribution, metabolism, or excretion of drugs.
* History of photosensitivity to quinolones.
* Use of systemic antibiotic within 30 days of screening.
* Confirmed lifetime history of C. difficile diarrhea
* History of spontaneous tendon rupture
* History of smoking or use of nicotine containing products within 3 months of screening or a positive urine cotinine indicative of smoking at screening.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams of alcohol: 12 fluid ounces (fl oz) (360 millilitre [mL]) of beer, 5 fl oz (150 mL) of wine, or 1.5 fl oz (45 mL) of 80-proof distilled spirits.
* History of sensitivity to any of the study drugs or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK medical monitor, contraindicates the potential subject's participation.
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if the clinical research unit uses heparin to maintain IV cannula patency).
* A positive pre-study hepatitis B surface antigen or positive hepatitis C antibody result within 3 months of screening or positive human immunodeficiency virus (HIV) antibody.
* A positive urine test for drugs of abuse at screening or at Day -1; positive urine test for alcohol (or alcohol breath test) within 24 hours of any dose in the study.
* Exclusion criteria for screening and baseline ECG (a single repeat test is allowed for eligibility determination): Heart rate: <40 and >100 beats per minute (bpm) (For males), <45 and >100 bpm (For Females); PR interval<120 and >220 millisecond (msec); QRS duration<70 and >110 msec; QTcF interval>450 msec.
* Evidence of previous myocardial infarction (does not include ST-segment changes associated with repolarization).
* Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular block [second degree or higher], Wolff-Parkinson-White syndrome), sinus pauses >3 seconds, non-sustained or sustained ventricular tachycardia (>3 consecutive ventricular ectopic beats), or any significant arrhythmia that, in the opinion of the investigator and GSK medical monitor, will interfere with the safety of the individual subject.
* An abnormal finding of clinical significance in the arrhythmia detection Holter performed on Day -2, which in the view of the investigator would compromise subject safety or interfere with study procedures or assessments will be excluded from the study. Full disclosures will be reviewed in detail and the review maintained as part of the subject's source documents. Analysis of the Holter recordings will consider the following:
* Heart rate (significant brady- or tachycardia, based on investigator's judgment)
* Reports of symptomatic arrhythmia (except isolated extrasystoles)
* Normal and aberrant beats
* Number of supraventricular contractions, premature atrial contractions, premature ventricular contractions, couplets, triplets, and ventricular tachycardias
* Atrioventricular conduction defects
* Atrial fibrillation and flutter
* Participation in the study would result in a donation of blood or blood products in excess of 500 mL within a 56-day period.
* Participation in a clinical trial in which the subject has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2014-10-06 (Actual); Primary Completion 2015-03-02 (Actual); Study Completion 2015-03-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in corrected QT interval, using the Fridericia formula (QTcF) for GSK2140944 (1000 mg and 1800 mg) | Up to 48 hours
  ECGs will be measured using a 24-hour continuous 12-lead Holter monitor. ECGs will be extracted up to 10 replicates at the following time points: at 3 time points pre-dose (45, 30, and 15 minutes prior to starting the infusion) and 0.25, 0.5, 1.0, 1.5, 2.0 (end of infusion), 2.5, 3.0, 4.0, 6.0, 8.0, 12.0, 24 and 48 hours after dosing, for a total of 16 time points per treatment period

SECONDARY OUTCOMES:
Change from baseline in ECG parameters for GSK2140944 (1000 mg and 1800 mg) | Up to 48 hours
  ECGs will be measured using a 24-hour continuous 12-lead Holter monitor at predefined timepoints. ECG parameters includes QT (QT interval), QT corrected according to the Bazett formula (QTcB), QT/RR pairs from the defined time points at which subjects are supinely resting (QTci), Individually corrected QT interval (QTcI), heart rate (HR), PR interval, and the complex of 3 of the graphical deflections seen on a typical ECG (QRS) interval
Categorical outliers in ECG parameters for GSK2140944 (1000 mg and 1800 mg) | Up to 48 hours
  ECGs will be measured using a 24-hour continuous 12-lead Holter monitor at predefined time points. Categorical outliers ECG parameters includes QTc, HR, PR, and QRS interval
Change from baseline in ECG parameters for moxifloxacin | Up to 48 hours
  ECGs will be measured using a 24-hour continuous 12-lead Holter monitor at predefined time points. ECG parameters includes QTcF, QTcB, QTci, QTcI, QT, HR, PR, and QRS interval
Composite of pharmacokinetic (PK) parameters for GSK2140944 (1000 mg and 1800 mg) | Up to 48 hours
  PK parameters including area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0-infinity]), area under the concentration-time curve from time zero (pre-dose) to time of last quantifiable concentration (AUC[0-t]), systemic clearance of parent drug (CL), maximum observed concentration (Cmax)
Composite of PK parameters for moxifloxacin | Up to 48 hours
  PK parameters including AUC(0-infinity), AUC(0-t), CL, apparent clearance of parent drug after oral dosing (CL/F), Cmax, λz, t1/2, tmax, Vss, Vz, apparent volume of distribution after oral dosing (Vz/F).
Plasma concentrations and change in QTcF for GSK2140944 and moxifloxacin | Up to 48 hours
  The relationship between GSK2140944 plasma concentration following single IV administration and the baseline adjusted QTcF interval corrected for placebo will be explored
Amount excreted (Ae) in urine of unchanged GSK2140944 (1000 mg and 1800 mg) | Up to 48 hours
  Urinary recovery of unchanged drug that is total amount of drug excreted in urine (Ae), calculated by adding all the fractions of drug collected over all the allotted time intervals
Fraction of the dose (fe) excreted in urine | Up to 48 hours
  Fraction of the dose (fe) will be calculated as, percentage fe= (Ae/Dose) × 100
Renal clearance | Up to 48 hours
  Renal clearance of drug will be calculated as: Ae/ AUC(0-t)
Assessment of ECG | Up to Day 48
  Single 12-lead safety ECGs will be obtained at predefined time points using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals
Change from baseline in vital sign measurements | Up to Day 48
  Vital signs includes temperature, systolic and diastolic blood pressure and pulse rate and respiratory rate
Number of subjects with adverse events (AEs) | Up to Day 48
  An AE is any untoward medical occurrence in a subject or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Toxicity grading of clinical laboratory test results | Up to Day 48
  Clinical laboratory parameters includes hematology, clinical chemistry, and urinalysis

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Hossain M, Zhou M, Tiffany C, Dumont E, Darpo B. A Phase I, Randomized, Double-Blinded, Placebo- and Moxifloxacin-Controlled, Four-Period Crossover Study To Evaluate the Effect of Gepotidacin on Cardiac Conduction as Assessed by 12-Lead Electrocardiogram in Healthy Volunteers. Antimicrob Agents Chemother. 2017 Apr 24;61(5):e02385-16. doi: 10.1128/AAC.02385-16. Print 2017 May. PMID 28223381
- See also: Results for study 115775 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/115775?search=study&b'search_terms=115775'#rs
- Available data/document: Statistical Analysis Plan: 115775 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115775 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115775 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115775 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115775 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115775 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115775 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register